CLINICAL TRIAL: NCT02538393
Title: An Open Label, Randomized, Four-way Crossover Study in Healthy Male Subjects to Assess the Relative Bioavailability of Sorafenib Tablet for Oral Suspension Compared to Marketed Tablet and to Investigate the Pharmacokinetics of Sorafenib Tablet for Oral Suspension Including Food Effect and Dose Proportionality
Brief Title: Relative Bioavailability of Sorafenib Tablet for Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18175; 2015-002083-16 (EudraCT Number)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Biological Availability
MeSH Terms: interventions — Sorafenib; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A-C-B-D (Experimental): Subjects received a single oral dose of 400 mg sorafenib marketed tablets (2 * 200 mg) in fasting state (Treatment A) in the first intervention period; followed by a single oral dose of 200 mg sorafenib tablets for oral suspension (2 * 100 mg) in fasting state (Treatment C) in the second intervention period; followed by a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) in fasting state (Treatment B) in the third intervention period; and then a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) after a high-fat, high-calorie breakfast (fed state) (Treatment D) in the fourth intervention period. A washout period of at least 10 days was maintained between sorafenib administrations.
  Interventions: Drug: Sorafenib (BAY43-9006) Film-coated tablet; Drug: Sorafenib (BAY43-9006) Oral suspension
- Treatment B-A-D-C (Experimental): Subjects received a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) in fasting state (Treatment B) in the first intervention period; followed by a single oral dose of 400 mg sorafenib marketed tablets (2 * 200 mg) in fasting state (Treatment A) in the second intervention period; followed by a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) after a high-fat, high-calorie breakfast (fed state) (Treatment D) in the third intervention period; and then a single oral dose of 200 mg sorafenib tablets for oral suspension (2 * 100 mg) in fasting state (Treatment C) in the fourth intervention period. A washout period of at least 10 days was maintained between sorafenib administrations.
  Interventions: Drug: Sorafenib (BAY43-9006) Film-coated tablet; Drug: Sorafenib (BAY43-9006) Oral suspension
- Treatment C-D-A-B (Experimental): Subjects received a single oral dose of 200 mg sorafenib tablets for oral suspension (2 * 100 mg) in fasting state (Treatment C) in the first intervention period; followed by a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) after a high-fat, high-calorie breakfast (fed state) (Treatment D) in the second intervention period; followed by a single oral dose of 400 mg sorafenib marketed tablets (2 * 200 mg) in fasting state (Treatment A) in the third intervention period; and then a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) in fasting state (Treatment B) in the fourth intervention period. A washout period of at least 10 days was maintained between sorafenib administrations.
  Interventions: Drug: Sorafenib (BAY43-9006) Film-coated tablet; Drug: Sorafenib (BAY43-9006) Oral suspension
- Treatment D-B-C-A (Experimental): Subjects received a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) after a high-fat, high-calorie breakfast (fed state) (Treatment D) in the first intervention period; followed by a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) in fasting state (Treatment B) in the second intervention period; followed by a single oral dose of 200 mg sorafenib tablets for oral suspension (2 * 100 mg) in fasting state (Treatment C) in the third intervention period; and then a single oral dose of 400 mg sorafenib marketed tablets (2 * 200 mg) in fasting state (Treatment A) in the fourth intervention period. A washout period of at least 10 days was maintained between sorafenib administrations.
  Interventions: Drug: Sorafenib (BAY43-9006) Film-coated tablet; Drug: Sorafenib (BAY43-9006) Oral suspension

INTERVENTIONS:
Drug: Sorafenib (BAY43-9006) Film-coated tablet — Subjects received a single oral dose of 400 mg sorafenib marketed tablets (2 * 200 mg) in fasting state in Treatment A
Drug: Sorafenib (BAY43-9006) Oral suspension — Treatment C: Subjects received a single oral dose of 200 mg sorafenib tablets for oral suspension (2 * 100 mg) in fasting state in the second intervention period; Treatment B: Subjects received a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) in fasting state in the third intervention period; Treatment D: Subjects received a single oral dose of 400 mg sorafenib tablets for oral suspension (4 * 100 mg) after a high-fat, high-calorie breakfast (fed state) in the fourth intervention period.

SUMMARY:
The primary objective of the study is to

• Investigate the relative bioavailability of sorafenib as 400 mg (4 x 100 mg) tablet for oral suspension formulation in comparison to 400 mg (2 x 200 mg) marketed tablet formulation.

The secondary objectives of this study are to

* Evaluate the dose proportionality in sorafenib pharmacokinetics for sorafenib tablet for oral suspension formulation after administration of 200 mg (2 x 100 mg) and 400 mg (4 x 100 mg) dose of sorafenib in fasted state
* Evaluate the effect of food on the pharmacokinetics of the tablet for oral suspension formulation after administration of a single dose of 400 mg sorafenib (4 x 100mg)
* Evaluate the taste and palatability of sorafenib (both formulations)
* Assess the safety and tolerability of sorafenib tablet for oral suspension in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 (inclusive) and 45 years (inclusive) at the first screening visit.
* Body mass index (BMI) between 18.0 (inclusive) and 32.0 kg / m² (inclusive).
* Non-smoker or former smoker who has stopped smoking at least 3 months before the first study drug administration
* Ability to understand and follow study-related instructions
* Any subject who is a sexually active man and has not been surgically sterilized must consent to use a condom during intercourse and ensure that his female partner practices adequate contraception, or he must be willing to refrain from sexual intercourse from the beginning of the trial until 30 days after last study drug administration.

Exclusion Criteria:

* Medical and surgical history:

  * Failure of a major organ system or a medical disorder that would impair the subject's ability to complete the study or that would alter the absorption and pharmacokinetics of the study drug
  * Active infections or other medical, psychological or social problems of sufficient severity to limit full compliance with the trial
  * Known severe allergies, non-allergic drug reactions, or multiple drug allergies
  * History of clinically significant metabolic, renal, hepatic, or cardiovascular disease or central nervous system disorder
  * Clinically significant illness within 30 days before first study drug administration.
  * Febrile illness within 1 week before the first study drug administration
  * Known hypersensitivity to study drug
  * Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Electrocardiogram (ECG), blood pressure, heart rate:

  * Clinically relevant findings in the ECG (e.g. a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTc-interval over 450 msec)
* Laboratory examination:

  * Clinically relevant deviations of the screened laboratory parameters from reference ranges (especially for gamma-GT, ALT, AST, or bilirubin)
  * Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Last Data Point Greater Than Lower Limit of Quantitation (LLOQ) of Sorafenib in Plasma (AUC[0-tlast]) After Single Oral Dose | Pre-dose (0 hour) to 120 hours post-dose
  Area under the concentration versus time curve from zero to the last data point greater than LLOQ after single dose of sorafenib were measured. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration After Single Dose Administration (Cmax) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Maximum observed drug concentration after single dose administration of sorafenib in plasma was measured. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration After Single Dose Administration Divided by Dose (Cmax/D) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Maximum observed drug concentration after single dose administration divided by dose of sorafenib in plasma was measured. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity After Single Dose (AUC) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Area under the concentration versus time curve from zero to infinity after single dose of sorafenib in plasma was measured. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity After Single Dose Divided by Dose (AUC/D) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Area under the concentration versus time curve from zero to infinity after single dose divided by dose of sorafenib in plasma. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Last Data Point Divided by Dose (AUC[0-tlast]/D) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Area under the concentration versus time curve from zero to last data point divided by dose of sorafenib in plasma was measured. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Total Body Clearance of Sorafenib Calculated After Extravascular Administration (CL/F) | Pre-dose (0 hour) to 120 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time to Reach Maximum Concentration (tmax) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Time to reach maximum concentration of sorafenib in plasma.
Half-life Associated With the Terminal Slope (t1/2) of Sorafenib in Plasma | Pre-dose (0 hour) to 120 hours post-dose
  Half-life associated with the terminal slope of sorafenib in plasma. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Number of Subjects With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | From start of study treatment up to 30 days after the last sorafenib dose administration
  An adverse event (AE) was any untoward medical occurrence in subject who received study drug without regard to possibility of causal relationship. AEs that started or worsened after first administration of study medication up to 30 days after end of treatment with study medication were considered to be treatment-emergent (TE). A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly and another medical important serious event as judged by investigator. SAEs that started or worsened after study drug treatment were recorded as TESAEs.
Number of Subjects With Various Acceptance Regarding the Taste and Palatability of the Tablet Formulations | Within 5 to 10 min of each administration of sorafenib
  For each administration of sorafenib, subjects completed a questionnaire regarding the taste and palatability of the tablets for oral suspension or marketed tablets within 5 to 10 min after administration. Results from the questionnaire regarding the taste of tablet, aftertaste and overall impression of the two different tablet formulations were analysed. CD= Completely disagree; SD= Somewhat disagree; Ne= Neutral; SA= Somewhat agree; CA= Completely agree; Un= Unknown.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, Germany